CLINICAL TRIAL: NCT05895721
Title: A Randomized Control Trial of the Use of Virtual Reality as an Adjunct in the Treatment for Generalized Anxiety Disorders
Brief Title: Virtual Reality for Generalized Anxiety Disorders
Acronym: VR-GAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinical Research Centre, Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMRR-22-00741-C75
Record Dates: First submitted 2023-05-12; First posted 2023-06-09 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2023-09

CONDITIONS: Generalized Anxiety Disorder
Keywords: GAD; VR
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard Of Care only
- Intervention (Other): Standard Of Care + VR Modules
  Interventions: Other: Virtual Reality

INTERVENTIONS:
Other: Virtual Reality — Virtual Reality as adjunct treatment
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to apply Virtual Reality as an adjunct treatment for Generalized Anxiety Disorder. The main question it aims to answer are:

* Determination of the efficacy of VR modules as an adjunct therapy in improving GAD-7 scores
* Assessment of the acceptability of VR modules as an adjunct therapy to the standard of care

Participants will randomized into two arms:

* Control Arm: Standard of Care only
* Intervention Arm: Standard of Care + VR Modules

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-59
2. The primary diagnosis is a generalized anxiety disorder
3. Agree to participate and consented as per study protocol.
4. There is no change in the standard of care within the past two months prior to enrollment into the study. If a patient is on any psychotherapy, then there is no change in the type of current psychotherapy intervention.
5. GAD- 7 more than or equal to 5.
6. Able to come for the session as per scheduled.

Exclusion Criteria:

1. Documented or known case of permanent hearing/visual impairment e.g., vestibular abnormalities that represent significant contraindications for the use of VR or visual impairment e.g., cataract.
2. Documented Disorder as listed:

   * A. Psychosis
   * B. Psychosis disorder - previous case, known case of
   * C. Claustrophobia
   * D. Substance use
   * E. Personality disorder
   * F. Visual impairment that might hinder usage of virtual reality equipment
   * G. Intellectual disabilities
   * H. All types of seizures including febrile seizure
3. The patient is under more than 1 center during follow up (e.g., patient is also receiving treatment from a private hospital for GAD).

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
To determine the efficacy of VR modules as an adjunct therapy in improving GAD-7 scores among patients with generalized anxiety disorders. | Week 0 - Week 4
  Patient will be access with GAD-7 questionnaire repeatedly at different time interval (3 Times - Week 0, Week 2, Week 4) .

SECONDARY OUTCOMES:
To assess the acceptability of VR modules as an adjunct therapy to the standard of care among patients with generalized anxiety disorders. | Week 0 - Week 4
  Patient will assess with standard questionnaire on acceptability of VR technology (3 Times - Week 0, Week 2, Week 4).

CONTACTS AND LOCATIONS:
Locations (5):
- Malaysia (5):
  - Hospital Sultanah Aminah, Johor Bahru, Johor
  - Hospital Permai, Johor Bahru, Johor
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Hospital Kulim, Kulim, Kedah
  - Hospital Sultanah Nur Zahirah, Kuala Terengganu, Terengganu